CLINICAL TRIAL: NCT05973851
Title: A Randomised, Controlled Trial to Investigate the Effect of a Sixweek Intensified Pharmacological Treatment for Major Depressive Disorder Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Brief Title: The Effect of a Six Week Intensified Pharmacological Treatment for Major Depressive Disorder Compared to Treatment as Usual in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Acronym: INTENSIFY MDD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Inge Winter (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Sponsor-Investigator, Dr. Inge Winter, Principal Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-506617-21-00 (EU CT#)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Major Depressive Disorder; Treatment as usual; Early treatment-resistance
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Parallel randomization to the 2 arms, treatment as usual (TAU) or early-intensified pharmacological treatment (EIPT).
Who Masked: Outcomes Assessor
Masking Description: Open label, except for the assessors of the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray (Experimental): Major depressive disorder randomized to EIPT: Switch to second-line antidepressant + esketamine nasal spray or (es)ketamine infusion. Antidepressant: Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC).
  Esketamine nasal spray: 2 times per week for 4 weeks. Initial dose 28 mg, after that increases can be made with 28 mg per increase (up to 84 mg per week). This decision is up to the investigator's discretion (in accordance with SmPC).
  (Es)ketamine infusion: performed twice weekly for 4 weeks. Compound, brand up to the investigator's discretion (in accordance with SmPC).
  Interventions: Drug: Esketamine Nasal Product; Drug: Ketamine Hydrochloride; Drug: Esketamine hydrochloride
- Major Depressive Disorder TAU: second-line antidepressant (Active Comparator): Subject with major depressive disorder, randomized to TAU: switch to second-line antidepressant. When randomized to second-line anti-depressants, this means participants will receive treatment as usual. The physician has the choice to administer any second-line anti-depressant. More specification is not possible, as this is a choice the physician makes with the participant based on the characteristic and preference of the participant (in line with standard clinical practice).
  Interventions: Drug: Second-line Antidepressants

INTERVENTIONS:
Drug: Esketamine Nasal Product — See arm description
  Other Names: ATC code: N06AB10
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Ketamine Hydrochloride — See arm description
  Other Names: N01AX03
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Esketamine hydrochloride — See arm description
  Other Names: N015X14
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Second-line Antidepressants — See arm description
  Arms: Major Depressive Disorder TAU: second-line antidepressant

SUMMARY:
Over 28 million people suffer from current depressive disorder in the European Union. Major depressive disorder (MDD) is one of the most common psychiatric illnesses. The symptoms cause clinically significant distress or impairment in social, occupational, and other important areas of functioning. To treat MDD, there are several antidepressants available and prescribing medication is a process of trial-and-error. Guidelines do not explicitly advise on the order in which antidepressant medication should be prescribed. The choice of antidepressant should be tailored to the patient, while involving the patient in the decision-making process. In general, the choice for the first- and second-line treatment will be a second-generation antidepressant. Recently, esketamine nasal spray (intranasal (IN) administration) was approved for patients with treatment-resistant MDD (TRD). A patient is diagnosed with TRD when having used two antidepressants in sufficient duration and adequate dose without sufficient effect. TRD is associated with a negative impact on quality of life, higher risk for hospitalisations and suicide, comorbidities, poorer social and occupational functioning and a high carer burden. The efficacy of intranasal use of esketamine has been demonstrated in MDD subjects with treatment-resistant symptoms but also in subjects with non-treatment resistant depression, and is approved by the FDA and EMA as a third-line treatment. Besides the registered esketamine nasal spray, which is not available in all countries to all patients because of the high costs, off-label utilization of (es)ketamine infusions (IV) is growing extensively over time to treat TRD. Research conducted so far indicates an unequivocal initial substantial response to (es)ketamine IV in MDD populations, regardless of whether or not patients suffer from treatment resistant MDD. However, until now, there has not been a study investigating this in a sufficiently large population. This may be a unique opportunity to potentially prevent patients progressing into a treatment resistant illness stage. The potential implications of the results of the current study are the prevention of unnecessary trials of ineffective treatments, reducing subject burden substantially, as well as a reduction of healthcare and societal costs.

DETAILED DESCRIPTION:
Rationale Over 28 million people suffer from current depressive disorder in the European Union. Major depressive disorder (MDD) is one of the most common psychiatric illnesses. The symptoms cause clinically significant distress or impairment in social, occupational, and other important areas of functioning. To treat MDD, there are several antidepressants available and prescribing medication is a process of trial-and-error. Guidelines do not explicitly advise on the order in which antidepressant medication should be prescribed. The choice of antidepressant should be tailored to the patient, while involving the patient in the decision-making process. In general, the choice for the first- and second-line treatment will be a second-generation antidepressant. Recently, esketamine nasal spray (intranasal (IN) administration) was approved for patients with treatment-resistant MDD (TRD). A patient is diagnosed with TRD when having used two antidepressants in sufficient duration and adequate dose without sufficient effect. TRD is associated with a negative impact on quality of life, higher risk for hospitalisations and suicide, comorbidities, poorer social and occupational functioning and a high carer burden. The efficacy of intranasal use of esketamine has been demonstrated in MDD subjects with treatment-resistant symptoms but also in subjects with non-treatment resistant depression, and is approved by the FDA and EMA as a third-line treatment. Besides the registered esketamine nasal spray, which is not available in all countries to all patients because of the high costs, off-label utilization of (es)ketamine infusions (IV) is growing extensively over time to treat TRD. Research conducted so far indicates an unequivocal initial substantial response to (es)ketamine IV in MDD populations, regardless of whether or not patients suffer from treatment resistant MDD. However, until now, there has not been a study investigating this in a sufficiently large population. This may be a unique opportunity to potentially prevent patients progressing into a treatment resistant illness stage. The potential implications of the results of the current study are the prevention of unnecessary trials of ineffective treatments, reducing subject burden substantially, as well as a reduction of healthcare and societal costs.

Objective The primary objective is to compare the treatment response (baseline; visit 2 vs. end of treatment; visit 4), expressed as symptom severity at six weeks and changes in symptom severity from baseline, as measured through the Montgomery-Åsberg Depression Rating Scale (MADRS) under an early-intensified pharmacological treatment to that under treatment as usual, in subjects who had a first-time treatment failure of first-line treatment during the current episode of MDD.

Main trial endpoints Change in symptom severity total score from baseline (visit 2) to end of treatment (visit 4). This is measured using MADRS.

Secondary trial endpoints

1. To compare changes in severity and improvement in global functioning assessed by the Clinical Global Impression Scale (CGI) between the two treatment arms.
2. To compare changes in the levels of depression and anxiety between treatment arms.
3. To compare changes in quality of life and functioning measures between treatment arms.
4. To compare changes in cognitive performance between treatment arms.
5. To compare the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4.
6. To compare presence of side effects between treatment arms.
7. To compare use of concomitant medication between treatment arms.
8. To compare premature discontinuation (timing and reason) between treatment arms.
9. To compare changes in suicidal ideation between treatment arms.

Trial design The clinical study is an international, multicenter controlled, randomised, open label trial (with blinded raters), with a treatment duration of four weeks.

Trial population The aim is to recruit 418 subjects with major depressive disorder, without psychotic features. Male and female subjects, in- and out-patients, within the age range of 18 to 65 years old are eligible for participation. The main exclusion criteria are defined to protect the wellbeing of subjects, e.g. being pregnant or breastfeeding, subjects with previous failure on (es)ketamine, meeting any contraindications, or participants with a known intolerance to (es)ketamine.

Interventions

Subjects are randomised to treatment as usual (second-line treatment) or to the early-intensified pharmacological treatment (third-line treatment). Treatment per can be found in the table below:

Table 1. Overview of treatment randomisation per study sample. MDD sample Treatment as Usual (TAU) Switch to second-line antidepressant Early-Intensified Pharmacological Treatment (EIPT) Oral antidepressant plus esketamine nasal spray or esketamine IV or ketamine IV

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of subjects represented by the trial subjects as well as the nature and extent of burden and risks In the current study, clinical practice is mimicked as much as possible to maximize generalizability and for feasibility purposes. To this end, Summaries of Product Characteristics (SmPCs) are followed with regards to contraindications (implemented as exclusion criterion), safety measures and allowed combinations with other medications. Site visits and assessments are kept to a minimum to keep subject burden at an acceptable level, while meeting the objectives of the study. Blood samples for biomarker analyses are only collected when subjects provide consent; safety measures are performed as part of clinical routine.

Use of both EIPT and TAU medications implies that there is a risk of side effects. For TAU, these side effects are well-known, and would be no different from regular clinical practice. For EIPT, there are acute psychotropic effects of (es)ketamine which are considered side effects for this study, such as anxiety, delusional thoughts, dissociation and hallucinations (see IMPDs). In addition, increased blood pressure and heart rate, as well as dizziness and nausea are reported. These acute effect are transient and after 2 hours completely dissipated. Therefore, an observation period of 2 hours after every administration is implemented to monitor this closely. The potential side effects of all treatments are well-known and will be monitored during the study with a standardized side-effect scale (GASE), spontaneous reporting and the local standard procedure regarding other measures such as laboratory tests, physical examinations, ECGs. The results will be captured (as data) and reviewed for tolerability. Most of the tests that will be done as part of standard clinical care (lab tests, ECG, physical examination) for EIPT are also part of TAU.

A benefit of the study is that while ensuring that the tolerability and additional burden remains acceptable, the investigators expect that the larger effect in reducing symptom severity will justify the increase in burden relative to the TAU group. When participants are treated with the intense treatment in earlier stage of the illness (less trial and error before moving on to this treatment option), this is expected to result in a reduced burden of disease for subjects, expressed as less relapses, lower all-cause mortality, hospitalisations and job losses and improved quality of life, in addition to lower societal and healthcare costs as well as preventing patients from turning into a treatment-resistant treatment phase. Last, an advantage of participation could be that subjects will be more thoroughly followed and examined, and that therefore effects and side effects are measured and managed better.

IMPORTANT: the study was submitted to the European authorities before (see NCT05603104) and they requested to split this study into 3 studies (1 for each diagnostic category). The investigators have done this and created 3 new ClinicalTrials.gov studies as well, from which this is one for major depressive disorder. The ClinicalTrial.gov numbers for the other studies are NCT05958875 for INTENSIFY SZ and NCT05973786 for INTENSIFY BD. The site in the UK (London) followed the advice and will submit 3 separate protocols and are therefore included in the current record. However, Israel already submitted this as one protocol. Therefore, the investigators keep the old clinicaltrials.gov number for Israel (NCT05603104).

ELIGIBILITY:
Inclusion Criteria:

1. In- or outpatients, at least 18 years of age up until 65.
2. Being willing and able to provide written informed consent. Having a legal guardian to cosign is allowed. Informed consent will be signed at visit 1, before any study procedure.
3. Female subjects of child bearing potential must use effective contraception during the trial as per the requirements of the applicable SmPCs and should have a negative pregnancy test at visit 1 or 2 (before randomisation).
4. Meeting diagnostic criteria for a primary diagnosis of major depressive disorder (without psychotic features), according to DSM-5. The primary diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2).
5. Subject experiences a treatment failure due to lack of efficacy in the current episode, as confirmed by a CGI-I ≥3; perferably, this treatment is a first-line pharmacotherapeutic agent for the primary DSM-5 diagnosis, and was prescribed for at least 4 weeks within an effective dose range as specified in the Summary of Product Characteristics (SmPCs).
6. Subject and clinician intend to change pharmacotherapeutic treatment. However, other lines of treatment are allowed as well.
7. A minimum symptom severity threshold needs to be present (moderate level; see below) and subject needs to experience functional impairment.

   * The minimum symptom severity threshold is a score of ≥20 on the Montgomery Åsberg Depression Rating Scale (MADRS)
   * Functional impairment is defined as a score of 5 or higher on any of the three scales of the Sheehan Disability Scale (SDS).

Exclusion criteria:

1. Being pregnant or breastfeeding.
2. Subject has used (es)ketamine previously for the treatment of depressive symptoms.
3. Subject has a known intolerance to (es)ketamine or to all TAU medication.
4. Meeting any of the contraindications for (es)ketamine, or to all TAU medication options, as specified within the applicable SmPC, supported by clinically significant abnormal values on local laboratory tests, electrocardiogram (ECG) or physical examinations.
5. Subject has participated in another clinical trial in which the subject received an experimental or investigational drug or agent within 30 days before visit 1.
6. Subject experiences any other significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the trial, or may influence the result of the trial, or the subject's ability to participate in the trial.
7. Subjects with active suicidal ideation with some intent to act, without specific plan ("Yes" to question 4 of the Columbia-Suicide Severity Rating Scale (C-SSRS)) or active suicidal ideation with specific plan and intent ("Yes" to question 5 of the C-SSRS), followed by an assessment by the treating clinician who determines it is not safe for the subject to participate in the study
8. Subject meets criteria for current substance use disorder, as confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2). Nicotine dependency is allowed, as well as mild and moderate alcohol and/or cannabis use disorder (as defined by MINI v7.0.2). Severe alcohol and/or cannabis use disorder are not allowed.
9. Subjects have not been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
10. Subjects dependent on the sponsor, investigator or trial site must be excluded from participation in advance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the change in symptom severity on Montgomery Asberg Depression Rating Scale | 6 weeks
  Change in symptom severity (EIPT vs. TAU) total score from baseline (visit 2) to end of treatment (visit 4). This is measured using the Montgomery Asberg Depression Rating Scale. Minimum score is 0, maximum score 60. A bigger mean change means a better outcome

SECONDARY OUTCOMES:
Compare proportion of participants that is in symptomatic remission | 6 weeks
  Comparison of the proportion of participants (EIPT vs. TAU) that is in symptomatic remission at visit 4. Remission is defined as a Montgomery Asberg Depression Rating scale score of ≤ 12.
Compare the change in the severity and improvement CGI-S sub-scores | 6 weeks
  To compare changes in the severity sub-score of the Clinical Global Impression Scale (CGI 2) between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4). Higher scores indicate higher illness severity. Minimum score: 1, maximum score: 7
Compare the change in the severity and improvement CGI-I sub-scores | 6 weeks
  To compare changes in the total improvement sub-score of the Clinical Global Impression Scale (CGI 2) between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4). A higher score means lower treatment improvement. Minimum score: 1, maximum score: 7
Compare the changes in the levels of depression and anxiety | 6 weeks
  To compare changes in the levels of depression and anxiety as assessed with the Hospital Anxiety and Depression Scale between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4). Lower scores mean less depression and anxiety.
To compare changes in cognitive performance as measured through the Trail Making Test | 6 weeks
  To compare changes in cognitive performance as measured through the Trail Making Test between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A lower time to complete the test means better cognitive performance.
To compare the changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test | 6 weeks
  To compare changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means better cognitive performance.
To compare the changes in subjective cognitive performance as measured through the Perceived Deficits Questionnaire | 6 weeks
  To compare changes in cognitive performance as measured through the Perceived Deficits Questionnaire between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means worse subjective cognitive performance.
To compare the changes in functioning on the Leuven Affective and Pleasure Scale | 6 weeks
  To compare changes in the functioning measure, Leuven Affective and Pleasure Scale, between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, Maximum score: 160
To compare the changes in functioning on the Sheehan Disability Scale | 6 weeks
  To comparechanges in the functioning measure,Sheehan Disability Scale, between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means worse functioning. Minimum score: 0, maximum score 30.
To compare the changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form | 6 weeks
  To compare changes in quality of life measure, Quality of Life Enjoyment and Satisfaction Questionnaire Short Form between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). A higher scores means better quality of life. Minimum score: 16, maximum score: 80.
To compare the changes of participants in quality of life measure, Quality of Life Scale -100, subscale inner tension | 6 weeks
  To compare changes in quality of life measure, Quality of Life Scale -100, subscale inner tension between the two treatment arms over the four weeks treatment period (visit 2 versus visit 4). This is a dichotomous scale (unsatisfactory or satisfactory). More 'satisfactory' answers means higher quality of life.
To compare the frequency of occurrence of side effects between the two treatment arms. | 6 weeks
  To compare presence of side effects as measured through General Assessment of Side Effects Scale and reported spontaneously between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4). Higher scores means more side effects. Minimum score: 0 side effects, maximum score: 38 side effects.
To compare the proportion of participants using concomitant medication between the two treatment arms. | 6 weeks
  To compare use of concomitant medication between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4) effects.
To compare the proportion of participants who prematurely discontinue between the two treatment arms. | 6 weeks
  To compare premature discontinuation between the two treatment arms (EIPT/TAU) over the four week treatment period (visit 2 versus visit 4).
To compare the reason of participants that prematurely treatment discontinue the study between the two treatment arms. | 6 weeks
  To compare the difference in reason of participants that prematurely discontinue the study treatment between the two treatment arms.
To compare changes in suicidal ideation between treatment arms. | 6 weeks.
  Changes on the Columbia-Suicide Severity Rating Scale (C-SSRS) throughout the study; EIPT vs TAU. Higher scores means higher suicidal ideation. The maximum score is 5.

CONTACTS AND LOCATIONS:
Locations (12):
- Medical University Innsbruck, Innsbruck, Austria
- Germany (4):
  - Universitätsklinik für Psychiatrie und Psychotherapie Bielefeld, Bielefeld
  - LWL-Klinik Dortmund, Bereich Forschung & Wissenschaft, Dortmund
  - University Hospital Frankfurt am Main - Goethe University, Frankfurt am Main
  - Westfälische Wilhelms-Universität Münster, Münster
- Eginition Hospital, department of psychiatry, Athens, Greece
- Italy (4):
  - Universita degli Studi di Brescia, Brescia
  - University of Cagliari, Cagliari
  - Università degli studi della Campania Luigi Vanvitelli, Naples
  - Azienda Ospedaliero-Universitaria "Città della Salute e della Scienza di Torino", Turin
- Fundació Clínic per a la Recerca Biomèdica, Barcelona, Spain
- King's College London, Psychiatry & Cognitive Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR